CLINICAL TRIAL: NCT01764126
Title: Safety and Immunogenicity of Pneumococcal Protein Vaccine (PPrV) in Healthy Adults, Toddlers and Infants in Bangladesh
Brief Title: Pneumococcal Protein Vaccine Safety and Immunogenicity Trial
Acronym: PPR02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-11023; U1111-1117-7316 (Other: Sanofi Pasteur)
Record Dates: First submitted 2012-03-16; First posted 2013-01-09 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2013-01

CONDITIONS: Adverse Effects
Keywords: Safety; immunogenicity; pneumococcal; protein; vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumococcal protein vaccine (Active Comparator): Pneumococcal protein vaccine
  Interventions: Drug: Pneumococcal protein vaccine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Pneumococcal protein vaccine

INTERVENTIONS:
Drug: Pneumococcal protein vaccine — One dose of 50 µg of each of three proteins with adjuvant (aluminium hydroxide) IM
  Other Names: pneumococcal common protein vaccine
Drug: Pneumococcal protein vaccine — Three doses, 4 weeks apart, of 10 µg of each of three proteins with adjuvant (aluminium hydroxide) IM
  Other Names: pneumococcal common protein vaccine
Drug: Pneumococcal protein vaccine — Three doses, 4 weeks apart, of 25 µg of each of three proteins with adjuvant (aluminium hydroxide) IM
  Other Names: pneumococcal common protein vaccine
Drug: Pneumococcal protein vaccine — Three doses, 4 weeks apart, of 25 µg of each of three proteins without adjuvant IM
  Other Names: pneumococcal common protein vaccine
Drug: Pneumococcal protein vaccine — Three doses, 4 weeks apart, of 50 µg of each of three proteins with adjuvant (aluminium hydroxide) IM
  Other Names: pneumococcal common protein vaccine

SUMMARY:
This is an observer-blind, randomised, vaccine-controlled, vaccine trial to determine the safety and immunogenicity of a pneumococcal protein vaccine. It will use an age step-down approach beginning with adults, then toddlers then infants, with data safety review at each stage before stepping down to the next age group. Adults and toddlers will receive the same dose of this three-protein (trivalent) vaccine (PcpA, PhtD, and PlyD1 proteins) at 50µg each. Infants will then be started at a low dose (10 µg), then medium dose (25µg) then high dose (50µg), with safety reviews at each stage before ascending to the next highest dose. Infants will also receive concomitant standard EPI childhood vaccines. Safety will be assessed by close monitoring beginning on the day of vaccination (day 0) and for the subsequent seven days, with recording of solicited and non-solicited adverse events. Immunogenicity will be assessed by specific antibody response to the three proteins. The study aims to recruit 280 study subjects across all age groups.

DETAILED DESCRIPTION:
This is a Phase I, single-center, randomized, placebo-controlled, step-down observer-blind study to assess the safety and immunogenicity of a single injection PPrV vaccine containing 50 µg of each protein (PcpA, PhtD and PlyD1) withadjuvant in healthy adults and toddlers, and of 3 injections in healthy infants (following the Expanded Program on Immunization [EPI] schedule) at 3 ascending dose levels (all adjuvanted 10, 25, and 50µg of each protein per dose level; with an additional un-adjuvanted formulation at 25 µg of each protein per dose level).

Overall, there will be 5 Cohorts. In Cohort I, adults will receive 1 injection of adjuvanted 50 µg PcpA, PhtD and PlyD1 PPrV vaccine (high dose) or placebo.

In Cohort II, toddlers will receive 1 injection of adjuvanted 50 µg PcpA, PhtD and PlyD1 PPrV vaccine or placebo.

In Cohorts III, IV and V, infants will receive 3 injections of one of the following PPrV vaccine formulations: adjuvanted 10 µg each PcpA, PhtD and PlyD1 (low dose), adjuvanted 25 µg each PcpA, PhtD and PlyD1 (middle dose), unadjuvanted 25 µg each PcpA, PhtD and PlyD1 (middle dose un-adjuvanted), or adjuvanted 50 µg each PcpA, PhtD and PlyD1 (high dose) or placebo, according to the EPI schedule (at 6 weeks, 10 weeks and 14 weeks), as well as concomitant applicable standard of care childhood vaccines ( Quinvaxem® [DTwP-HepB-Hib] vaccine, Bacillus Calmette-Guérin vaccine (BCG) (if not received at birth), and oral poliomyelitis vaccine [OPV]).

As a safety precaution, this trial will use a step-down approach for enrollment: for adults, 1 vaccination and acceptable review of safety data collected through Day 7 after injection, followed by enrollment of toddlers, 1 vaccination and acceptable review of safety data collected through Day 7 after injection, and then enrollment of infants (3 injections, EPI schedule). For infants, step-wise dose ascension is conditional upon acceptable safety reviews, which will be conducted after completion of the third vaccination of the EPI series at each dose level, using safety data collected through Day 7 after each of the vaccinations.

An Independent Data Monitoring Committee (IDMC) will be established for safety oversight of this study, for which a formal IDMC charter will be developed. For all safety reviews, blinded safety data will be provided to the Sponsor's Safety Management Team (SMT). The review will be performed by the SMT with presentation of findings, as per standard early safety review process, to the Sponsor's Safety Management Oversight Team (SMOT) in order to assess whether proceeding to the next ascending dose level is appropriate. The results will be communicated to the IDMC after each review. A formal IDMC review is proposed following completion of the Cohort II (toddler) safety review, prior to enrollment of Cohorts III, IV, and V (infants).

The study scheme is summarized in Figure 1, and details of safety reviews are described in the periodic safety data review (SDR) section. Electronic data capture (EDC) will be used for the collection of data generated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Acute or chronic condition that would interfere with the ability to complete the observation period
* Allergy to egg or other vaccine components
* Receipt of antibiotics
* Receipt of immune modulating or blood products
* Receipt of pneumococcal vaccine or concomitant participation in other vaccine or drug trials

Ages: 6 Weeks to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 30 days
  We will measure solicited and unsolicited adverse events for seven days from the day of vaccination, and serious adverse events for 30 days following vaccination.

SECONDARY OUTCOMES:
Immunogenicity | 30 days
  We will assess the antibody response using standard methods for each of the three proteins in the vaccine against a pre-vaccination baseline. For infants, this will be done with each of the three vaccine doses.

CONTACTS AND LOCATIONS:
Overall Officials: W. Abdullah Brooks, MD, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh